CLINICAL TRIAL: NCT00206960
Title: Effects of Classical and Atypical Antipsychotics on Dopamine Receptor Binding of 123I-epidepride, Cognition, Startle Response and Extrapyramidal Side-effects in Drug-naive First-episode Schizophrenic Patients
Brief Title: Dopaminergic, Functional, Structural, and Cognitive Disturbances in First-episode Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birte Glenthoj (Other)
Collaborators: University of Copenhagen (Other); Glostrup University Hospital, Copenhagen (Other); Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); The Danish Medical Research Council (Other); Copenhagen Hospital Corporation (Other); Janssen-Cilag Ltd. (Industry); The Novo Nordic Foundation (Other)
Responsible Party: Sponsor-Investigator, Birte Glenthoj, Professor of Psychopharmacology and Neuropsychiatry, Danish Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 363002; KF 01-078/97; KF 01-012/98; KF 11-057/99
Record Dates: First submitted 2005-09-10; First posted 2005-09-21 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Schizophrenia
Keywords: drug-naive; epidepride; single tomography; D2 receptor; information processing; PPI; antipsychotic treatment; MRI; fMRI; cognitive disturbances
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Clopenthixol; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: zuclopenthixol
- 2 (Active Comparator)
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: zuclopenthixol — Patients will be administered zuclopenthixol orally in doses between 4 -24 mg/day, depending on an effective reduction of symptoms
  Other Names: Cisordinol
  Arms: 1
Drug: risperidone — Patients will be administered risperidone orally in doses between 1-6 mg/day, depending on an effective reduction of symptoms
  Other Names: Risperdal
  Arms: 2

SUMMARY:
We wanted to compare dopamine D2 receptor activity, brain structure, brain function, sensory gating and cognition in neuroleptic-naive schizophrenic patients and matched healthy controls. Additionally, we wanted to examine the effects of 3 months of treatment with either low doses of a typical or an atypical antipsychotic compound on the same functions. The hypotheses were that schizophrenic patients suffered from disturbances in brain function and structure, information processing, and extrastriatal D2 receptor activity, and that these disturbances would be related to each other and to psychopathology. Additionally, we expected the atypical compound to have an effect on some of the disturbances in information processing, and that the atypical compound - in contrast to the typical drug - would show extrastriatal over striatal selectivity.

DETAILED DESCRIPTION:
31 neuroleptic-naive schizophrenic patients and 25 matched controls were recruited from the greater Copenhagen area. The patients were randomized to treatment with either low doses of the typical antipsychotic compound, zuclopenthixol, or the atypical drug, risperidone. Patients and controls were examined at base-line and patients were re-examined after 3 months of treatment.The study has resulted in two finish Ph.D. theses (Torben Mackeprang and Birgitte Fagerlund).

The data has in part been published in:

Mackeprang T, Tjelle Kristiansen K, Glenthoj B. Prepulse inhibition of the startle response in drug-naïve, first-episode schizophrenic patients before and after 3 months of treatment with a typical or an atypical antipsychotic drug. Biological Psychiatry 2002; 52(9): 863-873.

and

Fagerlund B, Mackeprang T, Gade A, Hemmingsen R, Glenthoj BY. Effects of Low-Dose Risperidone and Low-Dose Zuclopenthixol on Cognitive Functions in First-Episode Drug-Naïve Schizophrenic Patients. CNS Spectr. 2004; 9: 364-74.

and

Glenthoj BY, Mackeprang T, Svarer C, Rasmussen H, Pinborg L, Friberg L, Baaré W, Hemmingsen R, Videbæk C. Frontal dopamine D2/3 receptor binding in drug-naïve first-episode schizophrenic patients correlates with positive psychotic symptoms and gender. Biological Psychiatry 2006; in press. Mar 30; [Epub ahead of print]. PMID: 16784819 [PubMed - as supplied by publisher].

We are at present conducting a five-year follow-up study of the same cohort of patients and controls and plan a ten-year follow-up as well. The follow-up studies focus on brain structure (MRI), brain function, information processing, and psychopathology. We will correlate changes in structure and function to treatment, but no interventions (pharmacological or otherwise) are planned.

ELIGIBILITY:
Inclusion Criteria:

* For patients: Clinical diagnosis of schizophrenia.
* The controls were matched to the patients.

Exclusion Criteria:

* Patients: Previous antipsychotic treatment, patients who were compulsorily hospitalised or deemed in acute need of medication, mental retardation
* Controls: psychiatric diagnosis, psychiatric diagnosis in first-degree relatives, drug abuse, mental retardation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 1998-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
All examinations are done at baseline (patients and controls). In the patient group, they are repeated after 3 months of treatment | prospective
PANSS | prospective
SANS | prospective
SAPS | prospective
MRI | prospective
fMRI | prospective
startle response | prospective
PrePulse Inhibition of the startle response (PPI) | prospective
Cognition | prospective

SECONDARY OUTCOMES:
The cognitive test battery comprised tests from the Cambridge Neuropsychological Test Automated Battery (CANTAB) as well as paper-and-pencil cognitive tests. | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Birte Glenthoj, MD, DMSc, Study Director — University of Copenhagen, Psychiatric Center Glostrup, Ndr. Ringvej, DK-2600 Glostrup, Denmark
Locations (6):
- Denmark (6):
  - Neurobiology Research Unit, University of Copenhagen, Rigshospitalet, Copenhagen
  - Dept. of Nuclear Medicine, University of Copenhagen, Bispebjerg Hospital, Copenhagen NV
  - University of Copenhagen, Dept. F, Bispebjerg Hospital, Copenhagen NV
  - University of Copenhagen, Dept. of Psychiatry E, Bispebjerg Hospital, Copenhagen NV
  - Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychiatric Center Glostrup, Glostrup Municipality
  - Danish Research Center for Magnetic Resonance Imaging, Hvidovre Hospital, Hvidovre

REFERENCES:
- [Result] Mackeprang T, Kristiansen KT, Glenthoj BY. Effects of antipsychotics on prepulse inhibition of the startle response in drug-naive schizophrenic patients. Biol Psychiatry. 2002 Nov 1;52(9):863-73. doi: 10.1016/s0006-3223(02)01409-9. PMID 12399139
- [Result] Fagerlund B, Mackeprang T, Gade A, Glenthoj BY. Effects of low-dose risperidone and low-dose zuclopenthixol on cognitive functions in first-episode drug-naive schizophrenic patients. CNS Spectr. 2004 May;9(5):364-74. doi: 10.1017/s1092852900009354. PMID 15115949